CLINICAL TRIAL: NCT00330798
Title: A Comparison of Topical Nepafenac to Placebo in Corneal Epithelial Healing Times and Postoperative Pain Relief of Patients Status Post-Photorefractive Keratectomy: A Double-Masked Randomized Prospective Study
Brief Title: A Comparison of Topical Nepafenac to Placebo in Corneal Epithelial Healing Times and Postoperative Pain Relief
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: Matthew Caldwell (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20060020H
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-05

CONDITIONS: Photorefractive Keratectomy
Keywords: Photorefractive Keratectomy

ARMS (2):
- Nevanac (Experimental): One drop, three times daily, in the assigned eye for the first three postoperative days
  Interventions: Drug: nepafenac 0.1%
- Acular LS (Placebo Comparator): One drop, three times daily, in the assigned eye for the first three postoperative days
  Interventions: Other: ketorolac 0.4%

INTERVENTIONS:
Drug: nepafenac 0.1% — Nepafenac 0.1% randomly assigned to one eye, with ketorolac 0.4% in the fellow eye for contralateral post-surgical use.
  Arms: Nevanac
Other: ketorolac 0.4% — Keterolac 0.4% randomly assigned to one eye, with nepafenac 0.1% in the fellow eye for contralateral post-surgical use.
  Arms: Acular LS

SUMMARY:
The purpose of this study is to compare healing times and subjective pain level responses of nepafenac to placebo after photo refractive keratomileusis (PRK) surgery.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older with healthy ocular status and pre-operative refractive anisometropia of less than 2.000 diopters between eyes undergoing bilateral PRK surgery.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Those desiring PRK in only one eye, those in need of additional topical eye medications, those with history of drug/alcohol abuse, women breastfeeding or pregnant.
* Other protocol-defined exclusion criteria may apply.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Subjective pain | Day 5

SECONDARY OUTCOMES:
Rate of epithelial healing | Time to event

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Caldwell, Principal Investigator
Locations (1):
- Lackland Air Force Base, San Antonio, Texas, United States

REFERENCES:
- [Result] Caldwell M, Reilly C. Effects of topical nepafenac on corneal epithelial healing time and postoperative pain after PRK: a bilateral, prospective, randomized, masked trial. J Refract Surg. 2008 Apr;24(4):377-82. doi: 10.3928/1081597X-20080401-11. PMID 18500088